CLINICAL TRIAL: NCT01414829
Title: Efficacy of Gastric Biopsy for Culture and Antibiotic Sensitivity Assessment and Comparing of Different Methods for Helicobacter Pylori Disclosure
Brief Title: Efficacy of Gastric Biopsy for Culture and Antibiotic Sensitivity Assessment
Status: Withdrawn | Type: Observational
Why Stopped: difficulty in recruiting parients
Sponsor: The Baruch Padeh Medical Center, Poriya (Other Government)
Responsible Party: Paritsky Maya, Baruch Padeh MC
Other Study IDs: paritsky1.ct.il
Record Dates: First submitted 2011-08-10; First posted 2011-08-11 (Estimated); Last update posted 2012-12-04 (Estimated); Status verified 2012-12

CONDITIONS: Other Diseases or Conditions | Patient
Keywords: Peptic disease; Helicobacter pylori; Different methods
MeSH Terms: interventions — Gastroscopy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — gastric biopsies
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Gastroscopy — The reason for gastroscopy will be not related to the study

SUMMARY:
Gastric biopsies will be taken to compare different methods of H.pylori disclosure.Standard methods will be compared to culture.

ELIGIBILITY:
Inclusion Criteria:

* all referred for gastroscopy with clinical or endoscopic signs of peptic disease

Exclusion Criteria:

* coagulation disorders
* pregnant women

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patient referred for gastroscopy because of clinical reasons
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2011-08; Primary Completion 2012-01 (Estimated); Study Completion 2012-01

CONTACTS AND LOCATIONS:
Overall Officials: Maya PAritsky, MD, Principal Investigator — Baruch Padeh MC, Israel